CLINICAL TRIAL: NCT03348059
Title: Anti-E1E2 (D32.10 Epitope-binding) Antibodies Status Prior Therapy Favors Direct-acting Antiviral Treatment Efficacy
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CRC_GHN_2017_005
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Chronic Hepatitis c
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Direct-acting antiviral therapy — HCV patients received direct-acting antiviral treatment for 12 or 24 weeks

SUMMARY:
The hypothesis was to check whether baseline anti-E1E2 antibodies could predict virological outcome in Hepatitis C virus (HCV)-infected patients receiving direct-acting antiviral treatment

DETAILED DESCRIPTION:
Presence of anti-E1E2 antibodies was previously associated with spontaneous cure of hepatitis C virus (HCV). The hypothesis was to check whether baseline anti-E1E2 antibodies could predict virological outcome in HCV-infected patients receiving direct-acting antiviral treatment

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* HCV patients treated with direct-acting antiviral treatment
* Patients with a prior treatment blood sample
* Patients with sustained virological response or virological relapse

Exclusion Criteria:

* HIV or hepatitis B virus (HBV) coinfection

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hepatitis C virus (HCV)-infected patients treated with direct-acting antiviral treatment
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with positive anti-E1E2 antibody level at treatment initiation | Baseline (treatment initiation day)
  Anti-E1E2 antibody levels were determined using optical densities obtained after dilution of patients' serum samples at 1/250 and 1/500. Samples with anti-E1E2 levels above 950 (OD value× 1000) were considered positive

CONTACTS AND LOCATIONS:
Locations (1):
- Croix-Rousse Hospital, Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: No